**Official Title of the study:** Effectiveness of a Pre-procedural Mouthwash in Reducing Bacteria in Dental Aerosols and Splatters: a Randomized Clinical Trial

**Unique Protocol ID:** CAAE: 41244315.4.0000.5506

Date of the document: March 30, 2017

## STATISTICAL ANALYSIS

The total number of CFUs in the plates placed on the support board, clinician and volunteer, as well as all locations grouped were computed for each volunteer and then averaged in each group. For the support board, the mean number of CFUs of the three plates per volunteer was computed. For the Checkerboard DNA-DNA hybridization analysis, the mean levels of each bacterial species were averaged within each participant and then across participants in each of the four groups. After this, the percentage of the total DNA probe counts (proportions) was determined per volunteer and averaged across volunteers within each group. In addition, the proportions of the species belonging to the six complexes and the "other" group defined by Socransky et al.1998 were added to generate the proportion of each complex per group. The significance of differences between groups for the microbial data and for age were determined by Kruskall-Wallis and Dunn tests. Chi-square test was used to compare the differences in the frequency of gender and smoking status. The level of significance was set at 5%.